CLINICAL TRIAL: NCT06548685
Title: Vegetable Ivory Bone Material Study to Evaluate Whether a Biobased Natural Vegetable Ivory Formulation Can Produce Similar or Better Results Compared to Current Standard Bone Healing Treatments
Brief Title: Vegetable Ivory Bone Material in Bone Healing Compared to Current Standard Methods of Bone Healing
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mark Stanczyk (Industry)
Responsible Party: Sponsor-Investigator, Mark Stanczyk, VP, Dentivia, LLC
Organization: Dentivia, LLC (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Dentivia
Record Dates: First submitted 2024-07-23; First posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Bone Volume
Keywords: Vegetable Ivory Bone Material
MeSH Terms: interventions — Bone Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Participant 1 (Other): Bone grafting at one site and Vegetable Ivory Bone grafting at a parallel site in a tooth socket bone preservation intervention where the "drug' is the vegetable ivory bone replacement material in one site and human allograft bone graft on the other.
  Interventions: Procedure: Bone Grafting; Other: Vegetable Derived
- Participant 2 (Other): Bone grafting at one site and Vegetable Ivory Bone grafting at a parallel site in a tooth socket bone preservation intervention where the "drug' is the vegetable ivory bone replacement material in one site and human allograft bone graft on the other.
  Interventions: Procedure: Bone Grafting; Other: Vegetable Derived
- Participant 3 (Other): Bone grafting at one site and Vegetable Ivory Bone grafting at a parallel site in a tooth socket bone preservation intervention where the "drug' is the vegetable ivory bone replacement material in one site and human allograft bone graft on the other.
  Interventions: Procedure: Bone Grafting; Other: Vegetable Derived
- Participant 4 (Other): Bone grafting at one site and Vegetable Ivory Bone grafting at a parallel site in a tooth socket bone preservation intervention where the "drug' is the vegetable ivory bone replacement material in one site and human allograft bone graft on the other.
  Interventions: Procedure: Bone Grafting; Other: Vegetable Derived
- Participant 5 (Other): Bone grafting at one site and Vegetable Ivory Bone grafting at a parallel site in a tooth socket bone preservation intervention where the "drug' is the vegetable ivory bone replacement material in one site and human allograft bone graft on the other.
  Interventions: Procedure: Bone Grafting; Other: Vegetable Derived

INTERVENTIONS:
Procedure: Bone Grafting — Bone grafting in some sites and Vegetable Ivory Grafting in Parallel sites
Other: Vegetable Derived — Tooth extraction followed by socket preservation with vegetable ivory
  Other Names: Tooth socket preservation using Vegetable Ivory

SUMMARY:
The purpose of this research study is to evaluate whether a biobased natural vegetable ivory formulation can produce similar or better results compared to the current standard bone healing treatment.

DETAILED DESCRIPTION:
The patient is identified and surgical site and sides reviewed. The patient is consented to have bilateral tooth extractions which are mirror images of each other either in the maxilla or mandible.

Local anesthesia is administered and attention directed to the bilateral identified teeth. Each tooth is luxated with a straight elevator and removed with a forcep with out bony removal. The sites are curetted as indicated, irrigated with normal saline irrigation , then the sterile bone graft material (allograft and vegetable ivory bone graft) are reconstituted with sterile normal saline and placed in the tooth sockets then sutures with a 3-0 gut suture. Once hemostasis is obtained and pot operative care instructions are given, the patient is monitored for 30 minutes following the procedure then discharged.

ELIGIBILITY:
Inclusion Criteria:

Have parallel sites from which teeth have been extracted

Exclusion Criteria:

They are not a candidate for bone grafting or a dental implant

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Number of participants with completely healed bone graft surgical site | Six Months
  The number of participants who have bone volumes that match or exceed the control sites.

CONTACTS AND LOCATIONS:
Overall Officials: Pasquale Scutari, D.D.S., Principal Investigator — St Joseph's Hospital, Syracuse

IPD SHARING:
Plan to Share IPD: No